CLINICAL TRIAL: NCT07008911
Title: CardioHeartConnect: Commercially Available Fitness mHealth for Cardiac Rehabilitation Among Individuals Recovering From Transcatheter Aortic Valve Replacement
Brief Title: CardioHeartConnect: Commercially Available Fitness for Cardiac Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-0628; R61HL169336 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Disease
Keywords: Cardiac Rehabilitation; Transcatheter Aortic Valve Replacement; TAVR; Mobile Health; Peloton
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the exercise modules (intervention) group or the education only (control) group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CardioHeartConnect (CHC, Peloton Modules) (Experimental): Participants will receive access to an eight-week series of pre-set, clinically reviewed Peloton exercise modules delivered via the Ortus-iHealth platform. They will also receive a smartwatch designed to monitor physical activity and support engagement in cardiac rehabilitation after Transcatheter Aortic Valve Replacement (TAVR).
  Interventions: Behavioral: CardioHeartConnect
- CardioHeartEd (CHE, Informational Materials) (Active Comparator): Participants will receive access to an eight-week series of cardiac rehabilitation-related educational materials developed by the American College of Cardiology, delivered through the Ortus-iHealth platform. Participants in this arm will also receive a smartwatch to parallel the intervention group and support activity tracking.
  Interventions: Behavioral: CardioHeartEd

INTERVENTIONS:
Behavioral: CardioHeartConnect — Participants in the CardioHeartConnect group engage in an eight-week digital cardiac rehabilitation program using the commercially available Peloton app. The intervention includes two daily modules (10-25 minutes total) on weekdays, focused on walking, strength, low-intensity cardio, yoga, pilates, and stretching. Modules progress in intensity over time. The program is delivered through the Ortus-iHealth platform, which prompts daily participation and integrates survey responses and smartwatch data. The intervention is designed to support physical activity, functional capacity, quality of life, and cardiovascular health among patients recovering from Transcatheter Aortic Valve Replacement (TAVR).
  Other Names: CHC
  Arms: CardioHeartConnect (CHC, Peloton Modules)
Behavioral: CardioHeartEd — CardioHeartEd is the control condition in which participants receive weekly cardiac rehabilitation-related educational resources through the Ortus-iHealth platform for eight weeks. The content is created by the American College of Cardiology and is designed to promote cardiovascular health following TAVR. Participants also receive a smartwatch to wear for self-monitoring, but do not receive structured exercise content. The CHE group controls for access to technology and general education about heart health.
  Other Names: CHE
  Arms: CardioHeartEd (CHE, Informational Materials)

SUMMARY:
This trial evaluates the effectiveness of CardioHeartConnect, an eight-week mobile cardiac rehabilitation intervention using Peloton fitness modules, compared to educational control among patients recovering from transcatheter aortic valve replacement (TAVR). The study aims to improve physical activity, functional capacity, quality of life, and cardiovascular health using wearable devices and a digital engagement platform. A total of 200 patients will be recruited from the UCHealth Structural Heart and Valve Clinic and randomized to either CardioHeartConnect or CardioHeartEd. Participants will be assessed at baseline, 8 weeks, and 12 months using surveys, smartwatch data, and electronic health records.

DETAILED DESCRIPTION:
Despite strong evidence supporting cardiac rehabilitation (CR), participation following transcatheter aortic valve replacement (TAVR) remains low, particularly among patients with comorbidities, from underserved populations, or in rural areas. This randomized controlled trial tests the effectiveness and implementation of CardioHeartConnect (CHC), an eight-week, home-based cardiac rehabilitation intervention delivered through the commercially available Peloton app and supported by the Ortus-iHealth platform.

Two hundred patients recovering from TAVR at the UCHealth Structural Heart and Valve Clinic will be randomized 1:1 to either CardioHeartConnect or an attention control group, CardioHeartEd (CHE), which receives American College of Cardiology educational materials. All participants receive a smartwatch and access to the Ortus platform for data capture. CHC participants complete daily Peloton modules focusing on low-impact exercises including walking, stretching, yoga, and strength, tailored to CR guidelines and monitored by the research team.

The primary outcome is change in physical activity, measured by average daily steps at 8 weeks. Secondary outcomes include functional capacity (Duke Activity Status Index, VO2 max), cardiovascular health status (Life's Essential 8), health-related quality of life (Kansas City Cardiomyopathy Questionnaire), and self-efficacy. Safety events, participation in traditional CR, and implementation outcomes guided by the RE-AIM framework will also be assessed. Participants are followed for 12 months post-randomization.

This trial aims to inform scalable, equitable strategies for delivering CR through commercially available mobile health tools, particularly for patients who are underserved or waitlisted for traditional programs.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate for cardiac rehabilitation (CR) referral, as determined by the UCHealth Structural Heart & Valve Clinic team
* Community-dwelling
* Reside in the United States
* Able to speak and understand English
* Able to provide informed consent
* Able to stand with or without an assistive device
* Able to see and hear content on the Peloton App via phone, tablet, or computer

Exclusion Criteria:

- Determined to be inappropriate for cardiac rehabilitation referral by the UCHealth Structural Heart and Valve Clinic team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity measured by average daily steps | Baseline to 8 weeks (Primary); 8 weeks, and 12 months (Secondary)
  Change in mean daily steps from baseline to 8 weeks, measured using smartwatch accelerometer data collected through the Ortus platform. Steps will serve as the primary endpoint to evaluate the effect of CardioHeartConnect compared with control.

SECONDARY OUTCOMES:
Change in functional capacity (self report) | Baseline, 8 weeks, and 12 months
  Change in self-reported functional capacity measured by the Duke Activity Status Index (DASI) to assess physical function and cardiovascular fitness.
Changes in functional capacity (smart watch) | Baseline, 8 weeks, 12 months
  Estimated V02 max is generated with heart rate and motion data from smart watches. This is a measure of the maximum amount of oxygen your body can consume during exercise, useful for the very fit to those managing illness. A higher V02 max indicates a higher level of cardio fitness and endurance.
Change in cardiovascular-related quality of life | Baseline, 8 weeks, and 12 months
  Changes in Kansas City Cardiomyopathy Questionnaire (KCCQ) to assess symptom burden, well-being, and overall cardiovascular health.
Changes in cardiovascular health status | Baseline, 8 weeks, and 12 months
  Life's Essential 8 domains including diet, physical activity, nicotine exposure, sleep, BMI, blood pressure, cholesterol, and blood glucose.
Healthcare utilization | 8 weeks, 12 months
  Routine clinical visits, urgent care and emergency department visits, all cause hospitalizations
Changes in self-efficacy | Baselin, 8 weeks, 12 months
  Self-Efficacy for Managing Chronic Disease 6-item to assess ability to manage cardiovascular health.

OTHER OUTCOMES:
Safety tracking | 8 weeks and 12 months
  Injury from exercise and falls will be assessed using EHR including hospitalizations, emergency department visits, urgent care visits and mortality safety endpoints.
Participation in physical activity programing & cardiac rehab | 8 weeks and 12 months
  Self-report of participation in PA programming (i.e. silver sneakers); frequency Enrollment and attendance to usual CR
Intervention acceptability | 8 weeks
  Adapted user-rated mobile application rating scale for assing the acceptability and usabiltiy of digital tools.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Portz, PhD, MSW, Principal Investigator — University of Colorado, Denver; Christopher Knoepke, PhD, MSW, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth Structural Heart and Valve Clinic, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No